CLINICAL TRIAL: NCT01868997
Title: A Multicenter, Double-Masked, Placebo-Controlled, Efficacy And Safety Study Of RV 001, An Insulin-Like Growth Factor-1 Receptor (IGF-1R) Antagonist Antibody (Fully Human), Administered Every 3 Weeks (q3W) By Intravenous (IV) Infusion In Patients Suffering From Active Thyroid Eye Disease (TED)
Brief Title: Teprotumumab (RV 001) Treatment in Patients With Active Thyroid Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TED01RV; FD004792-01A1 (Other: FDA - Office of Orphan Product Development (OOPD)); 2014-000113-31 (EudraCT Number)
Record Dates: First submitted 2013-05-02; First posted 2013-06-05 (Estimated); Results first posted 2017-08-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Thyroid Associated Ophthalmopathies; Thyroid-Associated Ophthalmopathy
Keywords: Thyroid Eye Disease, Graves Orbitopathy, Thyroid Associated; Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy; Eye Diseases | interventions — teprotumumab; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): A placebo infusion (normal saline) administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions.
  Interventions: Drug: normal saline
- Teprotumumab (Experimental): Teprotumumab administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions. All participants start treatment at a dose of 10 mg/kg. At Week 3, the dose is escalated to 20 mg/kg and kept constant for the remainder of the study.
  Interventions: Drug: teprotumumab

INTERVENTIONS:
Drug: teprotumumab
  Other Names: RV 001; HZN-001
  Arms: Teprotumumab
Drug: normal saline
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the efficacy, safety, and tolerability of RV 001 (teprotumumab), a fully human anti-IGF1R antibody, administered q3W for 6 months, in comparison to placebo, in the treatment of participants suffering from active TED.

"Funding Source - FDA OOPD"

DETAILED DESCRIPTION:
Study with completed results acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves' disease associated with active TED and a clinical activity score of ≥ 4
* Fewer than 9 months from onset of TED
* No previous medical or surgical treatment, excluding local supportive measures and oral steroids if the maximum cumulative dose is less than 1000 mg methylprednisolone or equivalent with at least 6 weeks between last administration of oral steroids and randomization
* Euthyroid or with mild hypo or hyperthyroidism defined as free thyroxine (FT4) and free triiodothyronine (FT3) levels less than 50% above or below the normal limits (every effort should be made to correct the mild hypo- or hyperthyroidism promptly)

Exclusion Criteria:

* Optic neuropathy
* Corneal decompensation unresponsive to medical management
* Oral or IV steroid treatment for any non-TED reason in the preceding 3 months
* Poorly controlled diabetes
* Platelets < 100 x 10^9/L
* Hemoglobin concentration > 2 g/dL below the lower limit of normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2017-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (11):
  - Jules Stein Eye Institute at UCLA, Los Angeles, California
  - University of Denver, Aurora, Colorado
  - Emory University Department of Ophthalmology, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Department of Ophthalmology, Iowa City, Iowa
  - Kellogg Eye Center at University of Michigan, Ann Arbor, Michigan
  - Washington University Department of Ophthalmology, St Louis, Missouri
  - University of Nebraska Medical Center Department of Ophthalmology, Omaha, Nebraska
  - Casey Eye Institute at Oregon Health and Science University, Portland, Oregon
  - Hamilton Eye Institute at University of Tennessee, Memphis, Tennessee
  - Eye Wellness Center, Houston, Texas
  - Medical College of Wisconsin, The Eye Institute, Milwaukee, Wisconsin
- Johannes Gutenberg University Medical Center, Mainz, Germany
- Italy (2):
  - Fondazione Ca' Granda Ospedale Policlinico Graves GO Center, Milan
  - University of Pisa, Azienda Ospedaliera, Pisa
- Moorfields Eye Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Smith TJ, Kahaly GJ, Ezra DG, Fleming JC, Dailey RA, Tang RA, Harris GJ, Antonelli A, Salvi M, Goldberg RA, Gigantelli JW, Couch SM, Shriver EM, Hayek BR, Hink EM, Woodward RM, Gabriel K, Magni G, Douglas RS. Teprotumumab for Thyroid-Associated Ophthalmopathy. N Engl J Med. 2017 May 4;376(18):1748-1761. doi: 10.1056/NEJMoa1614949. PMID 28467880
- [Derived] Xin Y, Xu F, Gao Y, Bhatt N, Chamberlain J, Sile S, Hammel S, Holt RJ, Ramanathan S. Pharmacokinetics and Exposure-Response Relationship of Teprotumumab, an Insulin-Like Growth Factor-1 Receptor-Blocking Antibody, in Thyroid Eye Disease. Clin Pharmacokinet. 2021 Aug;60(8):1029-1040. doi: 10.1007/s40262-021-01003-3. Epub 2021 Mar 26. PMID 33768488
- [Derived] Wang Y, Smith TJ. Current concepts in the molecular pathogenesis of thyroid-associated ophthalmopathy. Invest Ophthalmol Vis Sci. 2014 Mar 20;55(3):1735-48. doi: 10.1167/iovs.14-14002. PMID 24651704

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 88 participants were enrolled (all participants who signed informed consent were considered enrolled in this study); 1 participant was never dosed and early terminated.
Groups:
- Placebo: A placebo infusion (normal saline) was administered once every 3 weeks (q3W) by intravenous (IV) infusion over a period of 24 weeks for a total of 8 infusions.
- Teprotumumab: Teprotumumab administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions. All participants started treatment at a dose of 10 mg/kg. At Week 3, the dose was escalated to 20 mg/kg and kept constant for the remainder of the study.
Period: Overall Study
Arm/Group | Placebo | Teprotumumab
Started | 45 (randomized and treated) | 42 (randomized and treated)
Completed | 38 | 36
Not Completed | 7 | 6
Not completed — Adverse Event | 2 | 5
Not completed — Lack of Efficacy | 2 | 0
Not completed — Other | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: A placebo infusion (normal saline) was administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions.
- Total: Total of all reporting groups
Arm/Group | Placebo | Teprotumumab | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (12.87) | 51.7 (10.78) | 52.9 (11.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 64
  Male | 9 | 14 | 23

OUTCOME MEASURES:

1. Primary Outcome: Responder Status at Week 24
Description: Number of participants classified as responders and non-responders at Week 24. Responders were defined as participants with a reduction in clinical activity score (CAS, see Outcome Measure 4 description for details) of ≥ 2 points, and a reduction in proptosis (amount of protrusion of the eye from the orbital rim) of ≥ 2 mm in the study eye, and no deterioration (increase in CAS of ≥ 2 points or increase in proptosis of ≥ 2 mm) in the non-study eye. Participants who had no assessment at 24 weeks were considered non-responders.
Time Frame: Week 24
Population: Intent to Treat Population: all participants who were randomized to treatment and received at least 1 dose of medication (either teprotumumab or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
Participants
  Responder | 9 | 29
  Non-Responder / Missing | 36 | 13
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p < 0.001, Regression, Logistic — Odds ratio, 95% confidence interval, and P-value are obtained from a logistic regression model with treatment and smoking status as covariates; Odds Ratio (OR) = 8.86, 95% CI 2-sided [3.293 to 23.825]

2. Secondary Outcome: Overall Average Change From Baseline in Graves' Ophthalmopathy Quality of Life (GO-QOL) Scale - Overall to Week 24 (Mixed-Model Repeated Measures [MMRM])
Description: The GO-QOL is a 16-item self-administered questionnaire used to assess the perceived effects of thyroid eye disorder (TED) by the participants on their daily physical and psychosocial functioning. Two subscales of the 16-question GO-QOL have been defined: Visual Functioning and Appearance, with 8 questions comprising each subscale. The transformed overall score is the sum of scores from all 16 questions to a scale of 0 (worst health) to 100 (best health).
Time Frame: Baseline to Week 24
Population: Intent to Treat Population: all participants who were randomized to treatment and received at least 1 dose of medication (either teprotumumab or placebo). A change from baseline of zero was imputed at the first postbaseline visit for participants with no postbaseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
units on a scale | 6.77 (2.251) | 17.74 (2.423)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p = 0.001, Mixed-Model Repeated Measures; Difference in Least Squares Mean = 10.97, 95% CI 2-sided [4.561 to 17.375], Standard Error of Mean 3.221

3. Secondary Outcome: Overall Average Change From Baseline in Proptosis of the Study Eye to Week 24 (MMRM)
Description: Proptosis is the amount of protrusion of the eye from the orbital rim. Measurements were recorded using the Hertel exophthalmometer. Participants with a decrease ≥ 2 mm were considered improving, those with an increase or decrease < 2 mm were considered remaining stable, and those with an increase ≥ 2 mm were considered worsening.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
mm | -0.15 (0.188) | -2.46 (0.200)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p < 0.001, Mixed-Model Repeated Measures; Difference in Least Squares Mean = -2.31, 95% CI 2-sided [-2.843 to -1.772], Standard Error of Mean 0.269

4. Secondary Outcome: Overall Average Change From Baseline in CAS to Week 24 (MMRM)
Description: The 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amended CAS was used to evaluate clinical activity. For each of the following items, one point is given: spontaneous orbital pain, gaze evoked orbital pain, eyelid swelling that is considered to be due to active (inflammatory phase) Graves' ophthalmopathy (GO), eyelid erythema, conjunctival redness that is considered to be due to active (inflammatory phase) GO, chemosis, and inflammation of caruncle or plica. The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
units on a scale | -1.85 (0.172) | -3.43 (0.181)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p < 0.001, Mixed-Model Repeated Measures; Difference in Least Squares Mean = -1.59, 95% CI 2-sided [-2.073 to -1.098], Standard Error of Mean 0.245

5. Secondary Outcome: Overall Average Change From Baseline in GO-QOL Scale - Visual Functioning to Week 24 (MMRM)
Description: The GO-QOL is a 16-item self-administered questionnaire used to assess the perceived effects of TED by the participants on their daily physical and psychosocial functioning. Two subscales of the 16-question GO-QOL have been defined: Visual Functioning and Appearance, with 8 questions comprising each subscale. Transformed Visual Functioning score is the sum of scores from following 8 questions to a scale of 0 (worst health) to 100 (best health): bicycling, driving, moving around the house, walking outdoors, reading, watching television (TV), hobby or pastime, feel hindered.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
units on a scale | 7.51 (2.646) | 21.67 (2.891)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p < 0.001, Mixed-Model Repeated Measures; Difference in Least Squares Mean = 14.16, 95% CI 2-sided [6.549 to 21.773], Standard Error of Mean 3.827

6. Secondary Outcome: Overall Average Change From Baseline in GO-QOL Scale - Appearance to Week 24 (MMRM)
Description: The GO-QOL is a 16-item self-administered questionnaire used to assess the perceived effects of TED by the participants on their daily physical and psychosocial functioning. Two subscales of the 16-question GO-QOL have been defined: Visual Functioning and Appearance, with 8 questions comprising each subscale. Transformed Appearance score is the sum of scores from the following 8 questions to a scale of 0 (worst health) to 100 (best health): feel appearance has changed, feel being stared at, feel people react unpleasantly, influence on self-confidence, feel socially isolated, influence on making friends, appear less often on photos, try to mask changes in appearance.
Time Frame: Baseline to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Teprotumumab
Number analyzed (Participants) | 45 | 42
units on a scale | 6.60 (2.656) | 12.92 (2.836)
Statistical Analysis 1: Comparison: Placebo vs Teprotumumab; Test type: Superiority; p = 0.101, Mixed-Model Repeated Measures; Difference in Least Squares Mean = 6.32, 95% CI 2-sided [-1.255 to 13.901], Standard Error of Mean 3.810

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: Treatment emergent adverse events (TEAEs) are presented, defined as events with onset at the time of or following the start of treatment with study drug or an event starting before the start of treatment but increasing in severity following the start of treatment.
Groups:
- Safety Population: Placebo: A placebo infusion (normal saline) was administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions.
  Safety Population: participants who received at least 1 dose of study treatment, grouped by treatment actually received.
- Safety Population: Teprotumumab: Teprotumumab administered q3W by IV infusion over a period of 24 weeks for a total of 8 infusions. All participants started treatment at a dose of 10 mg/kg. At Week 3, the dose was escalated to 20 mg/kg and kept constant for the remainder of the study.
  Safety Population: participants who received at least 1 dose of study treatment, grouped by treatment actually received.
Arm/Group | Safety Population: Placebo | Safety Population: Teprotumumab
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/43
Serious Adverse Events (participants affected / at risk) | 1/44 | 5/43
Other Adverse Events (participants affected / at risk) | 21/44 | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population: Placebo (N=44) | Safety Population: Teprotumumab (N=43)
Optic neuropathy (Eye disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Hashimoto's encephalopathy (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population: Placebo (N=44) | Safety Population: Teprotumumab (N=43)
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Nausea (Gastrointestinal disorders) | 4 | 8
Fatigue (General disorders) | 6 | 3
Upper respiratory tract infection (Infections and infestations) | 4 | 0
Weight decreased (Investigations) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 8
Dizziness (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 3
Paraesthesia (Nervous system disorders) | 0 | 3
Somnolence (Nervous system disorders) | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any Investigator/institution that plans on presenting or publishing results provide written notification of their request a minimum of 60 days prior to presentation or publication. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsors' Intellectual Property rights.